CLINICAL TRIAL: NCT03536312
Title: Treatment in Thoracic Aortic Aneurysm: Surgery vs Surveillance (TITAN:SvS)
Brief Title: Treatment in Thoracic Aortic Aneurysm: Surgery vs Surveillance
Acronym: TITAN:SvS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ottawa Heart Institute Research Corporation (Other)
Collaborators: University of Calgary (Other); University Health Network, Toronto (Other); Institut universitaire de cardiologie et de pneumologie de Québec, University Laval (Other); Hamilton General Hospital (Unknown); Montreal Heart Institute (Other); University of Pennsylvania (Other); Massachusetts General Hospital (Other); McGill (Unknown); University of Michigan (Other); Ohio State University (Other); Icahn School of Medicine at Mount Sinai (Other); Washington University School of Medicine (Other); University Hospitals Cleveland Medical Center (Other); University of Alberta (Other); Mayo Clinic (Other); Medical University of South Carolina (Other); Nova Scotia Health Authority (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other); Horizon Health Network (Other); The University of Texas Health Science Center, Houston (Other); San Francisco Veterans Affairs Medical Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 20180007-01H
Record Dates: First submitted 2018-04-18; First posted 2018-05-24 (Actual); Last update posted 2025-09-22 (Actual); Status verified 2025-09

CONDITIONS: Ascending Aortic Aneurysm Enlargement; Ascending Aorta Aneurysm
Keywords: Ascending Aorta Aneurysm; Aneurysm; Randomized Control Trial
MeSH Terms: conditions — Aneurysm, Ascending Aorta; Aneurysm

STUDY DESIGN:
Intervention Model Description: Patients between the age of 18 and 79 with an asymptomatic ascending aortic aneurysm between 5.0 cm and 5.4 cm in maximal diameter are entered into the randomization study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Surveillance Arm (No Intervention): Patients in the Non-Operative Registry will be followed in clinic annually with a CT scan to monitor the status of their ascending aortic aneurysm, until the end of the study, the occurrence of an aortic event, or death.
- Surgery/Treatment Arm (Other): Patients in the Operative Registry will have thoracic aortic surgery
  Interventions: Procedure: Thoracic Aortic Surgery

INTERVENTIONS:
Procedure: Thoracic Aortic Surgery — Thoracic aortic surgery to treat thoracic aortic aneurysm
  Arms: Surgery/Treatment Arm

SUMMARY:
The ascending aorta conducts blood from the heart to the rest of the body. The ascending aorta can become enlarged, and the risk of tearing and rupturing becomes higher with larger aorta. When the ascending aorta tears or ruptures, the risk dying is high even if surgery is done as soon as possible. Traditionally, when the ascending aorta gets above 5.5 cm, surgery is recommended to replace the aorta. However, this threshold is based relatively weak evidence, and sometimes patients with smaller aorta can tear or rupture. On the other hand, surgery carries its own risk as well. Since there are risk of waiting or doing surgery, there is currently no great support for either approach for patients with a smaller aorta. In the TITAN SvS trial, patients with an ascending aorta between 5.0 to 5.5 cm is assigned by chance to the early surgery group, in which they will undergo replacement of aorta, or the surveillance group, in which they will be closely monitored. The chance of dying or suffer tearing or rupture of aorta between the two groups will be compared. The result of the trial will guide future practice for patients with enlarged ascending aorta.

This is a prospective, multi-centre randomized control trial that compares the all-cause mortality, aneurysm-related aortic events, rate of stroke, and quality of life for those patients undergoing early elective ascending aortic surgery to those patients undergoing surveillance. Patients referred for an ascending aortic aneurysm that meets the inclusion criteria will be randomized to the early elective surgery group or the surveillance group. Recruitment will end when the desired sample size is reached, and the patients will be followed for a minimum 2-year period. The primary objective of the trial is to compare the composite outcome of the all-cause mortality and incidence of acute aortic events between surveillance and elective ascending aortic surgery for patients with degenerative or bicuspid valve-related ascending aortic aneurysm after 2 years of follow up. The hypothesis is that the early surgery group will have a significantly lower all-cause mortality and incidence of acute aortic events at 2 years of follow up compare to the surveillance group. The result of this trial will provide evidence based guidance in the appropriate management of ascending aortic aneurysm based on the size criteria, and establish a large database for future investigations.

DETAILED DESCRIPTION:
All patients referred electively to a participating investigator for the evaluation of their ascending aortic aneurysm will be screened for study eligibility. Patients between the age of 18 and 79 with an asymptomatic ascending aortic aneurysm between 5.0 cm and 5.4 cm in maximal diameter are entered into the randomization study. Patients with ascending aortic aneurysm with a diameter of 4.5 cm - 4.9 cm will be observed with serial CT, and will be considered for enrollment into the trial once the aneurysm reaches 5.0 cm.

When the patient is first assessed in clinic, a pre-randomization evaluation will be completed. Baseline information of the patient, including demographics, past medical history, family history, medications, smoking habits, and the characteristics of the aneurysm, is collected. Measurements including weight, height, heart rate, blood pressure in both arms, is recorded. Basic blood work, including hemoglobin, white cell count, platelets, electrolytes, creatinine, random blood sugar, HbA1c, and cholesterol profile is taken for analysis. An electrocardiograph, chest X-ray, and a CT scan from the surgeon's institution is also obtained. SF-36, the quality of life questionnaire, will be completed by the patient. Those patients that are suitable for the trial based on inclusion and exclusion criteria will then be randomized en-site through a computer-generated randomization program.

For the patients randomized to elective surgery group, the surgery is scheduled within 10-12 weeks of randomization. In the interim, the patient will be placed on maximal medical therapy for their aneurysm, including beta-blocker, statin, and blood pressure control, and the doses of these medication will be individualized based on each patient's own physiological response. The types of surgery (ascending aortic replacement, Bentall procedure, valve-sparing root replacement, etc.) will be at the discretion of the surgeon. The details of the surgery and the patient's course of postoperative hospital stay is recorded. The patient will be managed postoperatively according to routine hospital care. After discharge, patients will be seen at 1 months for their routine postoperative follow up, then annually counting from their index clinic visit before the surgery. At the first postoperative clinic visit, weight, height, heart rate, blood pressure in both arms, is recorded. Basic blood work, including hemoglobin, white cell count, platelets, electrolytes, creatinine is taken for analysis. An electrocardiograph and chest X-ray will be obtained. All subsequent clinic visits can be done in person or by phone conducted by a study coordinator. A CT scan will be obtained at all subsequent clinic visits. Mortality status and occurrence of acute aortic event or stroke in the previous year will be assessed at every annual clinic visit. Quality of life assessment by SF-36 questionnaire will be completed by the patient in person or by phone at 1 year and 2 years follow-up. Annual follow-up will continue until either the patient dies or the trial ends. Patients who are randomized to the surveillance group will be placed on maximal medical therapy for their aneurysm, including beta-blocker, statin, and blood pressure control. The doses of these medication will be individualized based on each patient's own physiological response. The patients will undergo a CT scan of the chest at the first clinic visit then annually for the duration of the study. All CTs will be uploaded to a core CT imaging lab where the image will be reviewed by a Radiologist. If the aneurysm grows beyond 5.5 cm or the patient develop symptoms, the surgeon will consider the patient for surgery. At all clinic visits, in addition to CT, weight, height, heart rate, blood pressure in both arms, an electrocardiograph, and a chest X-ray will be obtained. The surveillance visits continue until either the patient dies, the trial ends, or surgery is considered. If the patient is no longer considered a suitable candidate for surgery or refuse surgery, follow-up will continue, and the patient will no longer be a part of the trial and will only be registered in the side arm.

ELIGIBILITY:
Inclusion Criteria:

1. Patients between the age of 18 and 79 inclusive.
2. Ascending aortic aneurysm between 5.0cm and 5.4cm in maximal diameter as measured by CT with contrast.
3. Patients with ascending aortic aneurysm with a diameter of 4.5 cm - 4.9 cm will be observed with serial CT, and will be considered for enrollment into the trial once the aneurysm reaches 5.0 cm.

Exclusion Criteria:

1. Patients who refused to be randomized
2. Patients with symptomatic attributable to ascending aortic aneurysms
3. Patients who are unable to provide informed consents
4. Patients who are unable to attend for regular follow-up/ remain compliant with protocol
5. Previous cardiac surgery
6. Patients whose primary indication for cardiac surgery is non-AsAA related
7. Known AsAA expansion rate exceeding 0.5 cm/year during the past 5 years
8. Arch aneurysms with no ascending aorta involvement (no aneurysmal segments before the innominate artery)
9. Ascending aortic and arch aneurysm with descending thoracic aorta involvement
10. Patients with known connective tissue disease (E.g. Marfan syndrome, Loey-Dietz syndrome, Turner syndrome etc) syndrome, etc.)
11. Patients with possible genetic aortopathies (eg known family history of aortic aneurysms/premature aortic dissections/ruptures)
12. Patients with inflammatory arteritis (e.g. takayasu's arteritis, syphilitic arteritis, etc.)
13. Female patients who are pregnant or planning to become pregnant
14. Patients who have a history or presence of a medical condition or disease or psychiatric condition that in the investigator's assessment would render the subject ineligible for study participation.
15. Patients who, in the opinion of the investigator, are deemed unfit for surgery for reasons that may include:

    * Severe pulmonary disease
    * Cr = 250umol/L
    * Child Pugh Class B or C
    * NYHA III or IV
    * MI within the last 6 months
    * Major surgical procedure or angioplasty within 3 months
    * Expected survival less than 5 years because of other disease (e.g. invasive cancer)

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 610 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2035-05-31 (Estimated); Study Completion 2035-05-31 (Estimated)

PRIMARY OUTCOMES:
All-cause mortality and incidence of acute aortic events in both surveillance and elective ascending aortic surgery groups for patients with degenerative or bicuspid valve-related ascending aortic aneurysm after 2 years of follow up. | 2 years
  At 2 years follow up, number of patients in surveillance versus treatment group suffering from mortality or acute aortic dissection

SECONDARY OUTCOMES:
Intraoperative mortality and 30 day mortality of ascending aortic aneurysm repair | 30 days from surgery
  Document death during surgery or within 30 days post surgery
Incidence of need for elective ascending aortic aneurysm repair in the surveillance group | 2 years
  How many patients on the surveillance arm of the trial need to have surgery prior to the end of trial surveillance
Non aneurysm related death | 2 years
  How many patients in either surgical or surveillance arm have a non aneurysm related death
Aneurysm related death | 2 years
  How many patients in either the surveillance or surgical arm have an aneurysm related death
Incidence of cerebrovascular accidents (CVA) | 2 years
  How many patients have a CVA on the surgical or surveillance arm
Annual growth rate in diameter of ascending aortic aneurysm in the surveillance group | 2 years
  Prospective assessment of the rate of growth in mm/yr of moderate sized ascending aortic aneurysms
Quality of life at 1 year and 2 years for both groups | 2 years
  Patients will fill in questionnaires to assess impact of surveillance strategy versus surgery on quality of life

CONTACTS AND LOCATIONS:
Overall Officials: Munir Boodhwani, MD, Principal Investigator — Ottawa Heart Institute Research Corporation; Jehangir Appoo, MD, Principal Investigator — University of Calgary
Locations (28):
- United States (15):
  - University of California at San Francisco Medical Center, San Francisco, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - University of Michigan, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - The Valley Hospital, Inc, Ridgewood, New Jersey
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Duke University, Durham, North Carolina
  - University Hospitals Cleveland, Cleveland, Ohio
  - Ohio State University Medical Center, Columbus, Ohio
  - The Trustees of the University of Pennsylvania, Philadelphia, Pennsylvania
  - MUSC Health University Medical Center, Charleston, South Carolina
  - University of Texas Health Science Centre, Houston, Texas
  - Baylor Scott & White Research Institute, Plano, Texas
- Canada (13):
  - University of Calgary, Calgary, Alberta
  - Mazankowski Alberta Heart Institute, Edmonton, Alberta
  - Horizon Health Network, Saint John, New Brunswick
  - Nova Scotia Health Authority, Halifax, Nova Scotia
  - Health Sciences North, Greater Sudbury, Ontario
  - Hamilton General Hospital, Hamilton, Ontario
  - London Health Sciences Centre, London, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Toronto General Hospital, Toronto, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - McGill University Health Centre, Montreal, Quebec
  - Institut universitaire de cardiologie et de pneumologie de Québec, Québec, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Guo MH, Appoo JJ, Wells GA, Chu M, Ouzounian M, Fortier J, Boodhwani M. Protocol for a randomised controlled trial for Treatment in Thoracic Aortic Aneurysm: Surgery versus Surveillance (TITAN: SvS). BMJ Open. 2021 May 26;11(5):e052070. doi: 10.1136/bmjopen-2021-052070. PMID 34039580